CLINICAL TRIAL: NCT00409760
Title: A Randomized, Double-blind, Multicenter, Multifactorial, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Valsartan and Amlodipine Combined and Alone in Hypertensive Patients.
Brief Title: Safety and Efficacy of Valsartan and Amlodipine Combined and Alone in Patients With Hypertension.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAA489A2201
Record Dates: First submitted 2006-12-07; First posted 2006-12-11 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
Keywords: HYEPRTENSION, VALSARTAN, AMLODIPINE, high blood pressure
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Amlodipine

INTERVENTIONS:
Drug: valsartan+amlodipine combination, valsartan, amlodipine

SUMMARY:
This trial will compare valsartan and amlodipine combination therapies to both valsartan and amlodipine, and placebo for the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients 18 years and older.
* Male or female patients are eligible.
* Female patients must be either post-menopausal for one year or surgically sterile, or using effective contraceptive methods such as barrier method with spermicide or an intra-uterine device. Hormonal contraceptive use is disallowed.
* Patients with mild to moderate essential diastolic hypertension (grades 1 and 2 WHO classification) measured by calibrated standard sphygmomanometer.
* Patients must have a MSDBP >= 90 mmHg and < 110 mmHg at Visit 1 (week -2 to -4), and a MSDBP >= 95 mmHg and < 110 mmHg at Visit 2 (week 0).
* Patients must have an absolute difference of =< 10 mmHg in their average sitting diastolic blood pressure between Visits 1 and 2.
* Patients who are eligible and able to participate in the study, and who consent to do so after the purpose and nature of the investigation has been clearly explained to them (written informed consent).

Exclusion Criteria:

* Severe hypertension (grade 3 WHO classification; MSDBP >=110 mmHg diastolic and/or MSSBP >= 180 mmHg systolic).
* Inability to discontinue all prior anti-hypertensive medications safely for a period of 14 weeks).
* Known Keith-Wagener grade III or IV hypertensive retinopathy.
* History of hypertensive encephalopathy or cerebrovascular accident at anytime prior to Visit 1 (week -2 to -4).
* Transient ischemic cerebral attack during the last 12 months prior to Visit 1 (week -2 to -4).
* Evidence of a secondary form of hypertension, such as coarctation of the aorta, hyperaldosteronism, unilateral renal artery stenosis, or pheochromocytoma, etc.
* Type 1 Diabetes Mellitus.
* Type 2 Diabetes Mellitus with poor glucose control as defined by fasting glycosylated hemoglobin (HbA1c) >8% at Visit 1 (week -2 to -4).
* Administration of any agent indicated for the treatment of hypertension within a minimum 4 weeks prior to randomization into the study (Visit 2, week 0), with the permitted exception of those anti-hypertensive medications requiring tapering down commencing at Visit 0 (week -4 to -6).
* Known or suspected contraindications, including history of allergy to angiotensin receptor blockers or calcium channel blockers.
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1930 (Actual)
Dates: Start 2003-01; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Visit 2) in mean sitting diastolic blood pressure at trough (Wk 4 and Wk 8)

SECONDARY OUTCOMES:
Change from baseline (Visit 2) in mean sitting systolic blood pressure at trough (Wk 4 and Wk 8)
Change from baseline (Visit 2) in standing diastolic and systolic blood pressure at trough(Wk 4 and Wk 8)
Sitting and standing pulse

CONTACTS AND LOCATIONS:
Overall Officials: Novartis pharmaceuticals, Study Chair — Sponsor GmbH
Locations (1):
- Sites in Germany, Multiple Locations, Germany

REFERENCES:
- See also: NOVARTIS PATIENT RECRUITMENT WEBSITE — http://www.novartisclinicaltrials.com/webapp/etrials/home.do